CLINICAL TRIAL: NCT03020121
Title: Validation of BD Onclarity™ HPV Assay With PreservCyt® -ASCUS Samples
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower than anticipated rate of subject enrollment
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BDS-USHPVPC-AC
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Uterine Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Colposcopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BD HPV assay on Viper LT (Experimental): The BD HPV specimen will be tested with the BD HPV assay on the Viper LT instrument. The results will be compared to adjudicated histology. A portion of the specimens will be compared to a composite comparator generated by results of both Digene HPV and a polymerase chain reaction (PCR) sequencing test.
  Device: BD HPV assay on Viper LT The BD HPV specimen will be tested with the BD HPV assay on the Viper LT instrument. The results will be compared to adjudicated histology. A portion of the specimens will be compared to a composite comparator generated by results of both Digene HPV and a polymerase chain reaction (PCR) sequencing test. Colposcopy/biopsy will be performed on all subjects.
  Interventions: Procedure: Colposcopy/biopsy

INTERVENTIONS:
Procedure: Colposcopy/biopsy — Colposcopy/biopsy will be performed on all subjects

SUMMARY:
The purpose of the study is to compare the results of the Becton Dickinson (BD) Human Papilloma Virus (HPV) Assay on the Viper LT instrument from Liquid-based cytology media diluted in HPV diluent to adjudicated histology results from biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Females who are greater than or equal to 21 years of age,
* Subjects with a ASCUS (Atypical Squamous Cells - Undetermined Significance) cytology result,
* Females who provide informed consent

Exclusion Criteria:

* Known pregnant
* Prior complete or partial hysterectomy involving removal of cervix
* Conization, LEEP, cervical laser surgery or cryosurgery on the cervix has been performed in the last twelve months
* Colposcopy clinic referral patients

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 18 months
  Sensitivity of the BD HPV Assay for the detection of cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN). Sensitivity is calculated: Number of subjects with a positive BD HPV test with adjudicated histology results of CIN2 or greater divided by the total number of subjects with adjudicated histology results of CIN2 or greater. Similar for CIN3 or greater.
Specificity | 18 months
  Specificity of the BD HPV Assay for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN). Specificity is calculated: Number of subjects with a negative BD HPV test with adjudicated histology results of less than CIN2 divided by the total number of subjects with adjudicated histology results of less than CIN2. Similar for CIN3 or greater.
PositivePredictive Value | 18 months
  Positive Predictive Value (PPV) of the BD HPV Assay for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN). Positive Predictive Value is calculated: Number of subjects with a positive result for the BD HPV test and adjudicated histology results of CIN2 or greater divided by the total number of subjects with positive result for the BD HPV test. Similar for CIN3 or greater.
Negative Predictive Value | 18 Months
  Negative Predictive Value (NPV) of the BD HPV Assay for detecting cervical disease as defined by Cervical Intraepithelial Neoplasia (CIN). Negative Predictive Value is calculated: Number of subjects with a negative result for the BD HPV test and histology results less than CIN2 divided by the total number of subjects with negative results for the BD HPV test. Similar for CIN3 or greater.
Likelyhood ratio | 18 months
  Likelihood ratio for the detection of cervical disease as defined by cervical intraepithelial neoplasia (CIN). The likelihood ratio for each BD HPV test outcome summarizes how many times more (or less) likely subjects with the disease (e.g. CIN2 or greater and CIN3 or greater) are to have that particular HPV test outcome than subjects without the disease.
Absolute Risk | 18 Months
  Absolute risk for the detection of cervical disease as defined by cervical intraepithelial neoplasia (CIN). The Absolute Risk (AR) of the disease(e.g., CIN2 or greater and CIN3 or greater) for each BD HPV test outcome is the probability of the disease for that particular BD HPV test outcome.
Relative Risk | 18 Months
  Relative Risk of the detection of cervical disease as defined by cervical intraepithelial neoplasia (CIN). Relative Risk is the ratio between two different absolute risks. The relative risk of having a disease (e.g., CIN2 or greater and CIN3 or greater), will be evaluated to compare two different BD HPV Assay test outcomes.
Positive Percent Agreement | 18 Months
  Positive percent agreement of the BD HPV Assay as compared to a composite HPV comparator incorporating results for the Digene Hybrid Capture 2 (HC2) HPV test and PCR/Sequencing on both strands of the PCR amplicon (bidirectional sequencing). Positive percent agreement is calculated: Number of subjects with a positive BD HPV test with composite comparator positive divided by the total number of subjects with composite comparator positive.
Negative PercentAgreement | 18 months
  Negative percent agreement of the BD HPV Assay as compared to a composite HPV comparator incorporating results for the Digene HC2 HPV test and Polymerase Chain Reaction (PCR)/Sequencing on both strands of the PCR amplicon (bidirectional sequencing). Negative percent agreement is calculated: Number of subjects with a negative BD HPV test with composite comparator negative divided by the total number of subjects with composite comparator negative.
Non reportable rate | 18 months
  .Non-reportable rate of BD HPV test. Non-reportable rate is calculated as the number of non-reportable BD HPV test results divided by the total number of BD HPV test results

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - American Pathology Partners Inc., Denver, Colorado
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Indiana University, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - Transgenomics, Omaha, Nebraska
  - Southwest Womens Health, Albuquerque, New Mexico
  - Tricore Reference Lab, Albuquerque, New Mexico
  - Research Pathology Associates, LLC, Irvington, New York
  - Research Pathology Associates, Charlotte, North Carolina
  - Center for Disease Detection, San Antonio, Texas
- BioVision, Outremont, Quebec, Canada